CLINICAL TRIAL: NCT05590351
Title: Efficacy of Mobile Health Application in Promotion of Exclusive Breast Feeding and Young Child Feeding Practices in Pakistan: A Randomized Controlled Trial
Brief Title: Efficacy of Mobile Health Application in Promotion of Exclusive Breast Feeding and Young Child Feeding Practices in Pakistan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Rozina Nuruddin, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-3424-20757
Record Dates: First submitted 2022-10-12; First posted 2022-10-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Malnutrition, Infant; Malnutrition, Child
Keywords: infant & young child feeding practices; stunting; wasting
MeSH Terms: conditions — Infant Nutrition Disorders; Child Nutrition Disorders; Growth Disorders; Cachexia

STUDY DESIGN:
Intervention Model Description: m-health coaching application
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): m-health coaching application
  Interventions: Behavioral: First diet: m-health coaching application
- Standard of care (Active Comparator): Face to face counselling
  Interventions: Behavioral: Face to Face counselling

INTERVENTIONS:
Behavioral: First diet: m-health coaching application — Intervention for the study would comprise of a culturally appropriate m-health application called first diet. This application will be developed considering the perceptions, barriers and facilitators identified through formative research. Content of the messages would focus on breastfeeding, its importance and early initiation within one hour of birth, significance of first feed i.e. colostrum, importance of EBF from birth till 6 months, introduction of complementary feeding to 6-8 months old infants and appropriate YCFP. These messages would be drafted in the local preferable language assessed during formative research. The content of the messages would be translated and then back translated to ensure validity. These messages will be short, contextual and tailored according to the women's stage of gestation, delivery and infant's age
  Arms: Intervention
Behavioral: Face to Face counselling — Women randomly enrolled in the non-interventional group will receive face-face nutritional counseling instead of mobile application. Once enrolled in the group, Research Assistant (RA) will collect relevant details on the baseline questionnaire like intervention group but on a paper-based questionnaire. Women will be given first face-face counseling on the day of enrollment. The counseling sessions will coincide with the routine vaccination and growth monitoring schedule of the infant after women deliver
  Arms: Standard of care

SUMMARY:
Early life nutrition is the key modifiable determinant of child growth, development, survival and diseases of adult onset. Pakistan ranks highest for neonatal mortality rate (44.2/1000 live births (LBs)) globally. One third of under-five deaths (74.9/1000 LBs) are attributable to high prevalence of stunting (38%), underweight (23%) and wasting (7%), greatly related to feeding practices. Given the low prevalence of exclusively breast fed (EBF) (48%) and use of minimum acceptable diet (13%), mitigation of early life nutritional risk through promotion of EBF and Young Child Feeding Practices (YCFP) provides a critical window of opportunity for intervention. Secondary Care Hospitals (SCH) of the Aga Khan Health Services Pakistan provide essential maternal and child health services for low-middle income population. Babies born at these SCHs are followed up for vaccination, growth-monitoring and other services at the closely affiliated Family Health Centers (FHCs) run by Lady Health Visitors (LHVs). We aim to examine the effectiveness of a locally designed m-Health application for empowering mothers for child nutritional care as a potentially sustainable approach. The first six months of formative research would identify perceptions, barriers and facilitators for EBF and YCFP using self-determination behavioral theory, among multi-parous pregnant mothers enrolled at three SCHs of Karachi. A randomization trial would be conducted during next 18 months among near-term pregnant women who have access to smart-phones. A culturally appropriate mhealth application called first diet would be developed to provide personalized push messages delivered weekly by the LHVs. Non-intervention group will receive face-face nutritional counselling by the research staff at FHC following routine vaccination and growth-monitoring schedule. Mothers would followed-up from one month prior to expected delivery to child's first birthday. We expect 20% improvement in rates of EBF and YCFP with m-Health intervention. If proven effective, m-health would be incorporated in routine child care provision by LHVs.

DETAILED DESCRIPTION:
Every infant has the right to good nutrition. Early life nutrition is the key modifiable determinant of child growth, development, health, survival and chronic diseases of adult onset. The first year of infant's life provides a window of opportunity to improve health through adoption of recommended infant feeding practices. Breast milk is one of the first nutrition sources that a baby must be introduced to for optimum nutrition, health and growth. It is not only an important determinant of the nutritional status of the child but is also beneficial to strengthen the immune system of the baby and their sensory and cognitive development through creation of an intimate bond between the mother and her baby. Breast milk production and its consumption by the baby is also integral for the health of the mother, as it prevents the mother from ovarian and breast cancer and keeps her healthy for future pregnancies.

World Health Organization (WHO), therefore, recommends exclusive breastfeeding for up to 6 months and continued breastfeeding for at least 1 year for babies. Exclusive breast feeding is defined as 'infant receiving only breast milk without any food or drink, including water. Young Child Feeding Practices (YCFP) refers to the optimal feeding practices for a child aged between 6-12 months. This study aims to promote exclusive breastfeeding and young child feeding practices among women residing in the urban setup in the main city of Karachi, Pakistan, by the use of m-health intervention. WHO defines m-health as 'the use of mobile and wireless technologies to support the achievement of health objectives.

Pakistan is the sixth most populous country of the world. It is signatory to global agreement on reduction of under nutrition among children. Although, during the last decade (2011-18), proportion of underweight and stunted children has declined from 32% to 29%, and 44% to 40.2% respectively, proportion of wasting is showing an increasing trend from 15% to 17.7%. Further, the improvement achieved is not substantial. A quarter of newborns are born with low birth weight. Neonatal mortality rate (44.2/1000 live births (LBs) contributes 57% to the under-five mortality rate (74.9/1000 LBs) where breast feeding plays a crucial role for survival.

According to National Nutrition Survey 2018, only 48% of children under the age of 6 months are exclusively breast fed which is a suboptimal rise from 38% during 2012-13. The survey also highlighted that only 45.8% of infants were breastfed within 1 hour of birth. Likewise, only 35.9% of the infants between 6-8 months of age were weaned on age-appropriate complementary feeding, 14.2% receive minimum dietary diversity, 18.2% receive minimum meal frequency and 3.7% receive minimum acceptable diet. However, all these complementary feeding indicators are well below acceptable levels and are on decline compared to National Nutrition Survey 2011 except for dietary diversity. Below acceptable level of IYCF practices are found to be associated with maternal age, maternal illiteracy, unemployment, and poor household wealth status.

Province of Sindh has unsatisfactory infant and child nutritional indicators. Only 48% of mothers practice early initiation of breastfeeding within one hour of delivery while EBF is reported by 52.3% of the mothers. Similarly, only 43.5% of the children receive age-appropriate complementary feeding. Also, IYCF indicators of Sindh are poor compared to the other provinces of Pakistan. The proportions of children with minimum acceptable diet, minimum meal frequency and minimum dietary diversity are only 2.2%, 16.9% and 12.6% respectively and are lower than national estimates.

With the surge of technology use worldwide, the usage of mobile phone is also increasing in Pakistan. As per December 2019, there were 165 million cellular subscribers with 76 million 3G/4G users with smart phone penetration of 35.9% in Pakistan, though the usage is greater among males compared to females. Among women, 20% have access to a smartphone, 6% have a feature device while 23% have a basic mobile phone.

Mobile health (m-Health) has the potential to transform healthcare delivery by providing tailored and repeated information to individuals. Nowadays, a great bulk of the reproductive population has access to internet and socio media. Due to its increasing popularity, it bears the potential for delivery of intervention to a large number of people at a low cost.

However, such intervention has not been tested out in province of Sindh, in an urban setup where this technology use is increasing significantly over time. Hence, this study would be an important step in providing scientifically sound evidence to the limited pool of available literature on the effectiveness of m-Health interventions aimed at health care workers providing maternal and neonatal services in Low Middle Income Countries.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women in the third trimester at 36 +/- 1 week of gestation.
2. Planned to stay in their respective areas for at least 1 year after delivery
3. Planned to get the infant immunized from the respective FHC of the hospitals.
4. Have access to smart phones with internet connection.
5. Registered and planning to deliver to any of the Secondary Care Hospitals
6. Can read and write in local language (English and/or Urdu).
7. Consent to participate and remain in the study until 1 year of child age

Exclusion Criteria:

1. High-risk including maternal neurological/heart/ autoimmune/renal disease, preeclampsia, placenta previa, multiple gestations (twins/triplets), fetal structural/genetic anomalies, fetal growth restrictions, and birth trauma/requiring NICU admission.
2. Women who plan to move to different location after delivery

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females as this study require pregnant women
Enrollment: 300 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Exclusive Breast Feeding (EBF) | 1 year
  EBF up to 6 months of age defined as proportion of infants of 0-6 months of age who are fed exclusively with breast milk
Introduction of age appropiate solid, semi-solid or soft foods | 1 year
  Introduction of age appropiate solid, semi-solid or soft foods defined as the proportion of infants 6-8 months of age who receive solid, semi-solid or soft foods.

SECONDARY OUTCOMES:
Early Initiation of Breastfeeding (EIBF) | 1 year
  EIBF is defined as the proportion of children put to the breast within one hour of birth
Continued BF at 1 year | 1 year
  Continued BF at 1 year defined as the proportion of children 12 months of age who are still on breast milk.
Mean Duration of BF | 1 year
  Mean Duration of BF defined as average duration an infant is breastfed for 12 months.
Minimum Acceptable Diet | 1 year
  Minimum acceptable diet is a composite variable and would be based on meal frequency and dietary diversity.
Minimum Meal Frequency | 1 year
  Minimum Meal Frequency defined as the average number of daily meals for children 6-12 months of age, who receive solid, semi-solid, or soft foods Infant and young child feeding indicator
Minimum Dietary Diversity | 1 year
  Minimum dietary diversity is defined as the proportion of children 6-12 months of age who receive food from 4 or more food groups
Acute Respiratory Infection (ARI) | 1 year
  Acute respiratory Infection will be defined as short, rapid breathing that is chest-related and/or difficult breathing that is chest-related. Percentage of children up to 1 year of age with symptoms of ARI at any time in the last 2 weeks preceding the follow-up.
Acute Diarrhea | 1 Year
  Acute Diarrhea will be defined as the passage of three or more loose or liquid stools per day (or more frequent passage than is normal for the individual). The frequent passing of formed stools is not diarrhea, nor is the passing of loose, "pasty" stools by breastfed babies. Percentage of children up to 1 year of age with symptoms of diarrhea at any time in the last 2 weeks preceding the follow-up.
Visit to the Emergency room | 1 year
  Visit to the Emergency room will be defined as the infant brought to the emergency room for management of any acute illness in the past 2 weeks.
Hospitalization | 1 year
  Hospitalization will be defined as the infant admitted to the hospital for diagnosis or management of any acute illness in the past 2 weeks.
Stunting (height-for-age) | 1 year
  Stunting will be defined as Children whose height-for-age Z-score is below minus two standards deviations (-2 SD) from the median of the reference population
Wasting (weight-for-height) | 1 year
  Wasting will be defined as the children whose Z-score is below (-2 SD) from the median of the reference populations are considered thin (wasted), or acutely undernourished
Overweight (weight-for-height) | 1 year
  Children whose weight-for-height Z-score is more than 2 standard deviations (+2 SD) above the median of the reference population is considered overweight.
Underweight (weight-for-age) | 1 year
  Children whose weight-for-age Z-score is below (-2 SD) from the median of the reference population are classified as underweight.

CONTACTS AND LOCATIONS:
Overall Officials: Rozina Nuruddin, PhD, Principal Investigator — Agha Khan University
Locations (1):
- The Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Ariff S, Saddiq K, Khalid J, Sikanderali L, Tariq B, Shaheen F, Nawaz G, Habib A, Soofi SB. Determinants of infant and young complementary feeding practices among children 6-23 months of age in urban Pakistan: a multicenter longitudinal study. BMC Nutr. 2020 Dec 16;6(1):75. doi: 10.1186/s40795-020-00401-3. PMID 33323127
- [Background] Sesso R, Barreto GP, Neves J, Sawaya AL. Malnutrition is associated with increased blood pressure in childhood. Nephron Clin Pract. 2004;97(2):c61-6. doi: 10.1159/000078402. PMID 15218331
- [Background] Wang CJ, Chaovalit P, Pongnumkul S. A Breastfeed-Promoting Mobile App Intervention: Usability and Usefulness Study. JMIR Mhealth Uhealth. 2018 Jan 26;6(1):e27. doi: 10.2196/mhealth.8337. PMID 29374000
- [Background] Noh JW, Kim YM, Akram N, Yoo KB, Cheon J, Lee LJ, Kwon YD, Stekelenburg J. Factors Affecting Breastfeeding Practices in Sindh Province, Pakistan: A Secondary Analysis of Cross-Sectional Survey Data. Int J Environ Res Public Health. 2019 May 14;16(10):1689. doi: 10.3390/ijerph16101689. PMID 31091768
- [Background] Jiang H, Li M, Wen LM, Hu Q, Yang D, He G, Baur LA, Dibley MJ, Qian X. Effect of short message service on infant feeding practice: findings from a community-based study in Shanghai, China. JAMA Pediatr. 2014 May;168(5):471-8. doi: 10.1001/jamapediatrics.2014.58. PMID 24639004
- [Background] Akber S, Mahmood H, Fatima R, Wali A, Alam A, Sheraz SY, Yaqoob A, Najmi H, Abbasi S, Mahmood H, Dibley MJ, Hazir T. Effectiveness of a mobile health intervention on infant and young child feeding among children </= 24 months of age in rural Islamabad over six months duration. F1000Res. 2019 Apr 25;8:551. doi: 10.12688/f1000research.17037.3. eCollection 2019. PMID 31700614
- See also: WHO.int. 2020. Infant And Young Child Feeding — https://www.who.int/news-room/fact-sheets/detail/infant-and-young-child-feeding
- See also: The World Health Organization's infant feeding recommendation," World Health Organization — https://www.who.int/news-room/fact-sheets/detail/infant-and-young-child-feeding
- See also: Newborns: improving survival and well-being. (2020) — https://www.who.int/news-room/fact-sheets/detail/newborns-reducing-mortality
- See also: Only 15pc children in Pakistan receiving minimum acceptable diet — https://www.thenews.com.pk/print/368185-only-15pc-children-in-pakistan-receiving-minimum-acceptable-diet